CLINICAL TRIAL: NCT00876083
Title: Post-marketing Surveillance Study Ultravist®-IMAGE IoproMide (UltrAvist®) to Gain Further Information on Tolerability and Safety in X-ray Examination
Brief Title: PMS Study Ultravist-IMAGE, IoproMide (UltrAvist) to Gain Further Information on Tolerability and Safety in X-ray Examination
Acronym: IMAGE
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Global Medical Affairs Therapeutic Area Head, Bayer Schering Pharma AG
Other Study IDs: 14692; UV0701; 13422; 13421; 14480; 13276; 14336; 14181; 13602; 14243; 13275; 14180; 14338; 13859; 14376; 14337; 14245; 13212; 14526; 14527; 14528; 14586; 14661
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2011-02-28 (Estimated); Status verified 2011-02

CONDITIONS: Diagnostic Imaging
Keywords: Drug utilization review
MeSH Terms: interventions — iopromide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Ultravist (Iopromide, BAY86-4877)

INTERVENTIONS:
Drug: Ultravist (Iopromide, BAY86-4877) — Patients with indication for an X-ray examination and for whom the radiologist has decided to use the contrast medium Ultravist.

SUMMARY:
The purpose of this study is to obtain data on the safety and efficacy of Ultravist application in usual daily use.The radiologist will administer the contrast medium to the patient as he/she would have done without the study. No other examinations will be performed than would have been done routinely.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication for an X-ray examination and for whom the radiologist has decided to use the contrast medium Ultravist.

Exclusion Criteria:

* No exclusion criteria besides the contraindications for the use of Ultravist as mentioned in the product information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of female and male patients who require an X-ray examination with contrast enhancement. Physicians should consult the full prescribing information for Ultravist before enrolling patients and familiarize themselves with the safety information in the product package label.
Sampling Method: Non-Probability Sample
Enrollment: 44920 (Actual)
Dates: Start 2008-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events | During and after Ultravist application on the day of examination

SECONDARY OUTCOMES:
General contrast quality in the region of interest as assessed by physicians | On the day of examination

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (21):
- Many Locations, Bosnia and Herzegovina
- Many Locations, China
- Many Locations, Germany
- Many Locations, Hungary
- Many Locations, Indonesia
- Many Locations, Iran
- Many Locations, Italy
- Many Locations, Malaysia
- Many Locations, Moldova
- Many Locations, Pakistan
- Many Locations, Philippines
- Many Locations, Poland
- Many Locations, Romania
- Many Locations, Russia
- Many Locations, Saudi Arabia
- Many Locations, Singapore
- Many Locations, South Korea
- Many Locations, Taiwan
- Many Locations, Thailand
- Many Locations, Ukraine
- Many Locations, Vietnam